CLINICAL TRIAL: NCT01660750
Title: A Multi-Center Phase Ib, Open-Label, Dose-Finding Pilot Study to Evaluate the Combination of Carfilzomib and Cyclophosphamide With Dexamethasone Prior to ASCT in Patients With Transplant Eligible Newly Diagnosed Myeloma
Brief Title: A Safety Study of Carfilzomib, Cyclophosphamide & Dexamethasone Prior to ASCT in Patients With Newly Diagnosed Myeloma
Acronym: 11-MM-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Criterium, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMyC 11-MM-01; CAR-IST-520 (Other: Onyx Pharmaceuticals)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed multiple myeloma; transplant eligible multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib, Cyclophosphamide, Dexamethasone (Experimental): All eligible subjects will receive Carfilzomib, Cyclophosphamide, and Dexamethasone.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — IV over 30 minutes on Days 1,2,8,9,15, and 16 every 28 days
  Other Names: PR-171; Kyprolis
Drug: Cyclophosphamide — PO on days 1, 8, and 15 every 28 days
  Other Names: Cytoxan
Drug: Dexamethasone — 40 mg weekly PO or IV on Days 1, 8, 15, and 22, every 28 days.
  Other Names: Decadron

SUMMARY:
This is a dose finding pilot study to evaluate the safety and determine the maximum tolerated dose of the combination of carfilzomib and cyclophosphamide with dexamethasone (Car-Cy-Dex) prior to autologous stem cell transplant (ASCT) in patients with newly diagnosed transplant eligible multiple myeloma.

DETAILED DESCRIPTION:
This is a dose finding pilot study to evaluate the safety and determine the maximum tolerated dose of the combination of carfilzomib and cyclophosphamide with dexamethasone (Car-Cy-Dex) prior to autologous stem cell transplant (ASCT) in patients with newly diagnosed transplant eligible multiple myeloma. The study will also explore the efficacy of Car-Cy-Dex including overall response after induction therapy, overall response at 3 and 6 months post ASCT, and time to progression, progression free survival, and time to next therapy if it occurs within 6 months post ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Cytopathologically or histologically confirmed diagnosis of MM
* Measurable disease, as indicated by one or more of the following:
* Serum M-protein ≥ 1.0 g/dL
* Urine Bence Jones protein ≥ 200 mg/24 hr
* Elevated Free Light Chain as per the International Myeloma Working Group (IMWG) criteria
* Males and females ≥ 18 years of age
* Life expectancy of more than 5 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate hepatic function, with bilirubin < 2 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.5 times ULN
* Serum Creatinine Clearance(CrCl) ≥ 30 mL/min, either measured or calculated using a standard formula (e.g. Cockcroft and Gault)
* Additional Laboratory Requirements
* Absolute neutrophil count (ANC) ≥1.0 x 109/L
* Hemoglobin ≥8 g/dL [transfusion permitted]
* Platelet count ≥50.0 x 109/L
* Screening ANC should be independent of granulocyte-and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for at least 2 weeks
* Patients may receive RBC or platelet transfusions, if clinically indicated, in accordance with institutional guidelines
* Written informed consent in accordance with federal, local, and institutional guidelines
* Patients must agree to practice contraception
* Male patients must agree not to donate semen or sperm.

Exclusion Criteria:

* Patients with non-secretory or hyposecretory MM
* Prior treatment for MM (prior radiation therapy or dexamethasone up to 160 mg for spinal cord compression is allowed. Other limited field radiation involving ≤ 1/3 of the pelvic area is also allowed)
* Plasma cell leukemia
* Pregnant or lactating females
* Major surgery within 21 days prior to first dose
* Congestive heart failure (CHF) (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction in the previous six months
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 14 days prior to first dose
* Patients receiving active treatment or intervention for any other malignancy or patients who, at the Investigator's discretion, may require active treatment or intervention for any other malignancy within 8 months of starting study treatment.
* Serious psychiatric or medical conditions that could interfere with treatment
* Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose and/or within 14 days before study treatment
* Contraindication to any of the required concomitant drugs, including antiviral (e.g. Valacyclovir) and proton-pump inhibitor (e.g. lansoprazole). Corticosteroid therapy in a dose equivalent to dexamethasone ≥ 1.5 mg/day or prednisone ≥ 10 mg/day. (Steroid use is allowed if necessary to treat spinal cord compression and/or hypocalcaemia.)
* Patients in whom the required program of oral and IV fluid hydration is contraindicated, e.g. due to pre-existing pulmonary, cardiac, or renal impairment
* Patients with primary systemic amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events as a measure of safety and tolerability | Throughout treatment, estimated to be 4-6 months per patients
  Review of adverse events for safety and to determine the maximum tolerated dose of the combination treatment.

SECONDARY OUTCOMES:
Overall Response after induction therapy | Every 28 days during induction therapy, estimated to be 4-6 months
  Overall response (PR, VGPR, CR, sCR)
Overall Response post ASCT | 3 and 6 months post ASCT
  Overall Response (PR, VGPR, CR, sCR) at 3 and 6 months post ASCT.
Time to Progression | Througout treatment and 3 and 6 months post ASCT
  Time to progression will be noted if it occurs within 6 months post ASCT.
Progression Free Survival | up to 6 months post ASCT
Time to Next Therapy | up to 6 months post ASCT
  Time to Next Therapy if occurs within 6 months post ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Jatin Shah, MD, Principal Investigator — AMyC; Brian GM Durie, MD, Principal Investigator — AMyC
Locations (5):
- United States (5):
  - Samuel Oschin Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - University of Massachusettes Memorial, Worcester, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided